CLINICAL TRIAL: NCT07205458
Title: The Effect of Web-Based Breastfeeding Education Based on the Information-Motivation-Behavioral Skills Model on Fathers' Breastfeeding Support.( First-Time Fathers.)
Brief Title: The Effect of Web-Based Breastfeeding Education Based on Knowledge, Motivation, Behavioral Skills Model on Fathers' Breastfeeding Support
Acronym: Fathersupport
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, dilek menekşe, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIBU-SBF-DM-1
Record Dates: First submitted 2025-09-18; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Paternal Involvement in Breastfeeding; Parental Support for Breastfeeding
Keywords: Breastfeeding,Paternal support,Parental involvement,Exclusive breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Single-blind randomization will be provided in the study to be conducted in first-time fathers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMB Model Web-Based Breastfeeding Education Group (Experimental): Fathers in this group will participate in a structured web-based breastfeeding education program based on the Information-Motivation-Behavioral Skills (IMB) Model during the first two weeks postpartum, followed by two motivational interview sessions. The program will be completed within two weeks after baseline assessment and will continue until postpartum day 42. Motivational interviews will begin between days 13-17 postpartum, with a second interview between days 21-30 postpartum, depending on fathers' needs. The intervention aims to improve fathers' breastfeeding knowledge, motivation, and supportive behaviors.
  Interventions: Behavioral: IMB Model Web-Based Breastfeeding Education Program; Behavioral: Motivational interview sessions, Breastfeeding self efficiay,Behavioral Skills
- Control Group (No Intervention): Fathers in the control group will be followed up according to routine hospital follow-up and breastfeeding education practices. They will receive standard postpartum care, which may include general breastfeeding information from healthcare providers. This process will continue until postpartum day 42. Structured web-based education or motivational interview sessions will not be provided. At the end of the study, families may access the web-based education if they wish.

INTERVENTIONS:
Behavioral: IMB Model Web-Based Breastfeeding Education Program — A structured, model-based online education program designed to increase fathers' knowledge about breastfeeding through interactive lessons, videos, and resources. Fathers will be informed about breastfeeding during the postpartum period. The breastfeeding knowledge test will be completed two weeks after baseline data collection, and motivational interviews will be planned according to fathers' needs.
  Other Names: Breastfeeding Support Education, Behavior Change Education
  Arms: IMB Model Web-Based Breastfeeding Education Group
Behavioral: Motivational interview sessions, Breastfeeding self efficiay,Behavioral Skills — Motivational interview sessions aimed to strengthen fathers' motivation for breastfeeding and improve supportive behaviors. These sessions will begin between postpartum days 13-17 after the information phase is complete. The number of sessions will be based on fathers' needs (minimum of two and up to four). Each session's duration will follow the Turkish Ministry of Health's Postpartum Care Guide (2018). The second session will occur between postpartum days 21-30. After the motivational interviews are completed, fathers will have received information and motivation according to the Information-Motivation-Behavioral Skills (IMB) Model. Education and interview sessions will continue until postpartum day 42, shaped according to fathers' needs. At the end of all trainings, fathers are expected to have developed the skills to support mothers during breastfeeding and to have gained self-efficacy in the breastfeeding process
  Arms: IMB Model Web-Based Breastfeeding Education Group

SUMMARY:
Breast milk is a highly bioavailable, easily digestible, and miraculous food that meets all the nutrient, energy, and fluid needs of the baby for physical, mental, and psychological development. International health organizations emphasize that breastfeeding is the key to sustainable development and recommend exclusive breastfeeding for the first six months, followed by continued breastfeeding with complementary feeding for two years or longer. However, only a limited proportion of infants, both globally and in Turkey, are exclusively breastfed during the first six months, which remains below the targeted rates set within the scope of sustainable development goals. When the factors underlying mothers' discontinuation of breastfeeding are examined, many social, cultural, and psychological reasons are reported. One of these reasons is spousal/father support. In recent years, studies have focused on fathers to increase breastfeeding rates. In this direction, breastfeeding training based on the Knowledge-Motivation-Behavioral Skills (BMB) model, planned to be given to fathers to support the breastfeeding process and to accompany mothers and babies in breastfeeding, is of great importance. In the literature, no web-based online study was found to support fathers in the breastfeeding process based on the BMB model. The fact that the training is based on a theoretical model and planned to be web-based in terms of accessibility for fathers constitutes the original aspect of the study. The aim of this study was to examine the effect of web-based breastfeeding education, based on the Knowledge-Motivation-Behavioral Skills Model, on fathers' breastfeeding support.

DETAILED DESCRIPTION:
Breastfeeding plays a vital role in ensuring the healthy growth and development of infants. Breastfed children are more likely to survive and reach their full developmental potential. Breast milk supports not only the physical but also the cognitive and psychological development of the child, and it has been shown to reduce the risk of obesity later in life. Additionally, in low-income and developing countries, breastfeeding significantly contributes to the reduction of malnutrition, infectious diseases, and child mortality. Beyond its benefits for infants, breastfeeding also has long-term positive effects on maternal health. These benefits persist throughout the lives of both mother and child, making breastfeeding a crucial practice that should be actively promoted and supported. The World Health Organization has emphasized the significance of breastfeeding, recognizing it as a key driver of sustainable development. It is recommended to initiate breastfeeding within the first hour after birth, continue exclusive breastfeeding for the first six months, and maintain breastfeeding for two years or longer with complementary feeding. However, global breastfeeding rates remain below the target of 50% by 2025.

During this process, both national and international health authorities have emphasized that the perceptions and attitudes of family members-particularly fathers-toward breastfeeding significantly influence mothers' perspectives on breastfeeding. Paternal support for breastfeeding has been shown to contribute to improved breastfeeding outcomes, and fathers play a crucial role in promoting breastfeeding. Supportive and positive attitudes of fathers toward their partners influence maternal breastfeeding self-efficacy during the postpartum period. Increasing fathers' knowledge, self-efficacy, and involvement in breastfeeding-related interventions positively affects mothers' breastfeeding experiences. However, studies investigating paternal behavior during the breastfeeding period have revealed that many fathers lack sufficient knowledge about breastfeeding and breast milk. Moreover, they often do not fully understand the significance of breastfeeding for both maternal and infant health. Fathers have also reported uncertainty about how to support the breastfeeding process and expressed a desire for guidance on how to assist their partners.

Basing nursing practices on a specific theoretical model has been shown to positively influence both the quality of nursing care and overall health outcomes. In this context, a variety of models have been developed to facilitate health education, individual development, and behavioral change in health-related practices. One such model is the Information-Motivation-Behavioral Skills (IMB) Model. The IMB model was developed to understand the social and psychological factors that influence health-related behaviors. According to this model, once individuals are provided with accurate health information and sufficient motivation, they are more likely to acquire and adopt positive behavioral skills.

In this framework, encouraging fathers to actively participate in the breastfeeding process may extend breastfeeding duration and positively influence the breastfeeding experience. Such involvement can also enhance the relationships between father and infant, father and mother, and mother and infant. Applying the IMB model may help fathers develop appropriate, simple, and effective behavioral skills based on their own motivation. Moreover, these acquired behaviors are expected to be sustainable and impactful over time. Therefore, the aim of the proposed study is to examine the effect of a web-based breastfeeding education program-designed in accordance with the Information-Motivation-Behavioral Skills (IMB) Model-on paternal support for breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* • Fathers aged 19 and over

  * Becoming a nuclear family
  * Father can read and write Turkish
  * Father is open to communication and cooperative
  * Becoming a father for the first time
  * The father continues to live with his wife
  * Having a healthy and full-term baby
  * Not having any known medical/mental illness
  * Volunteering to participate in the research
  * Have access to the Internet, a computer or a smartphone

Exclusion Criteria:

* Fathers who refuse to participate in the research
* Mothers experiencing postpartum depression
* Fathers whose babies are hospitalized in the neonatal intensive care unit
* Fathers who have multiple or premature babies
* Fathers who do not speak Turkish and are not open to communication
* Presence of conditions that would contraindicate breastfeeding
* Babies without health issues requiring surgical treatment

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 68 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-02-10 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of knowledge about breastfeeding in the study and control groups | Baseline (before training) and Post-intervention (postpartum day 14)
  To assess the "knowledge" component of the Information-Motivation-Behavioral Skills (IMB) Model, the Breastfeeding Knowledge Test-Father Form (BKT-FF) developed by Buldum et al. (2024) will be used. This test consists of 38 items. Each correct answer is scored as "1.00," while incorrect or "I don't know" responses are scored as "0.00." Total scores range from 0.00 to 38.00, with higher scores indicating greater breastfeeding knowledge among fathers, whereas lower scores suggest insufficient knowledge.

SECONDARY OUTCOMES:
Evaluation of fathers' breastfeeding attitudes and participation in the study and control groups | Post-intervention (postpartum day 24)
  Fathers' Attitude and Participation in Breastfeeding Scale (F-BAPS): To assessthe "motivation" component of the Information-Motivation-Behavioral Skills Model,theFathers' Attitude and Participation in Breastfeeding Scale (FAPBS) willbe used FAPBS consists of two sections: "Fathers' Attitudes TowardBreastfeeding (FATB)" and "Fathers' Participation in Breastfeeding (FPB)",comprising a total of 28 items. Responses in FAPBS are evaluated usingfive-point Likert scale. Positive items about breastfeeding are scored as(1=Strongly disagree, 2=Disagree, 3=Undecided, 4=Agree and 5=Strongly agree)and negative items are scored in reverse order The total FATB score rangesfrom 14 to 70, with a cut-off score of 58. Scores ≥58 indicate a positive attitude, while scores <58 indicate a negative attitude toward breastfeeding.The total FPB score ranges from 14 to 70, with a cut-off score of 58.Scores≥58indicate good participation, while scores <58 indicate poor participation in the breastfeeding process
Evaluation of fathers' breastfeeding support in study and control groups | Difference between fathers' breastfeeding support status before and after the training-Post-intervention (postpartum day 42.)
  The Breastfeeding Father Support Scale will be used to evaluate the "behavioral skills" component of the model scale, which consists of 21 items, is designed to assess fathers' support for breastfeeding for those with infants aged 0-2 years. There are no reverse-coded items in the scale, and it is evaluated based on the average item score. Each item is rated on a Likert-type scale with the following points: 1 = Strongly Disagree, 2 = Disagree 3 = Sometimes, 4 = Agree, 5 = Strongly Agree. The minimum score that can be obtained from the scale is 21, and the maximum score is 105. A higher score indicates that the father provided more support to their partner during the breastfeeding period.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK MENEKŞE, Associate Professor, Study Director — SAKARYA ÜNİVERSİTESİ; Hilal BÜLBÜL, PhD Student, Principal Investigator — Sakarya University
Locations (1):
- Sakarya Üniversitesi, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gutin SA, Harper GW, Moshashane N, Ramontshonyana K, Stephenson R, Shade SB, Harries J, Mmeje O, Ramogola-Masire D, Morroni C. Relationship, partner factors and stigma are associated with safer conception information, motivation, and behavioral skills among women living with HIV in Botswana. BMC Public Health. 2021 Dec 8;21(1):2231. doi: 10.1186/s12889-021-12268-5. PMID 34879845
- [Background] Del Ciampo LA, Del Ciampo IRL. Breastfeeding and the Benefits of Lactation for Women's Health. Rev Bras Ginecol Obstet. 2018 Jun;40(6):354-359. doi: 10.1055/s-0038-1657766. Epub 2018 Jul 6. PMID 29980160
- [Background] Mangrio E, Persson K, Bramhagen AC. Sociodemographic, physical, mental and social factors in the cessation of breastfeeding before 6 months: a systematic review. Scand J Caring Sci. 2018 Jun;32(2):451-465. doi: 10.1111/scs.12489. Epub 2017 Jun 1. PMID 28569436
- [Background] Taspinar A, Coban A, Kucuk M, Sirin A. Fathers' knowledge about and attitudes towards breast feeding in Manisa, Turkey. Midwifery. 2013 Jun;29(6):653-60. doi: 10.1016/j.midw.2012.06.005. Epub 2012 Jul 25. PMID 22840976
- [Background] deMontigny F, Gervais C, Lariviere-Bastien D, St-Arneault K. The role of fathers during breastfeeding. Midwifery. 2018 Mar;58:6-12. doi: 10.1016/j.midw.2017.12.001. Epub 2017 Dec 6. PMID 29272696
- [Background] Bode L, Raman AS, Murch SH, Rollins NC, Gordon JI. Understanding the mother-breastmilk-infant "triad". Science. 2020 Mar 6;367(6482):1070-1072. doi: 10.1126/science.aaw6147. No abstract available. PMID 32139527
- [Background] Perez-Escamilla R, Tomori C, Hernandez-Cordero S, Baker P, Barros AJD, Begin F, Chapman DJ, Grummer-Strawn LM, McCoy D, Menon P, Ribeiro Neves PA, Piwoz E, Rollins N, Victora CG, Richter L; 2023 Lancet Breastfeeding Series Group. Breastfeeding: crucially important, but increasingly challenged in a market-driven world. Lancet. 2023 Feb 11;401(10375):472-485. doi: 10.1016/S0140-6736(22)01932-8. Epub 2023 Feb 7. PMID 36764313